CLINICAL TRIAL: NCT00696761
Title: The Long Term Effects of Alfuzosin(Xatral XL) in LUTS/BPH Patients: Evaluation of Voiding and Storage Function According to Bladder Outlet Obstruction Grade and Bladder Contractility
Brief Title: The Long Term Effects of Alfuzosin(Xatral XL) in Lower Urinary Tract Symptoms(LUTS)/BPH Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Soo Choo, urology department, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L9990
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: BPH
Keywords: LUTS; BPH; bladder outlet obstruction; bladder contractility
MeSH Terms: conditions — Urinary Bladder Neck Obstruction | interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- group1 (Active Comparator): Bladder outlet obstruction index(BOOI)≥ 20, Bladder contractility index(BCI)≥ 100 Alfuzosin was administered daily (10 mg) for 12 month.
  Interventions: Drug: Alfuzosin
- group2 (Active Comparator): BOOI≥ 20, BCI<100 Alfuzosin was administered daily (10 mg) for 12 month.
  Interventions: Drug: Alfuzosin
- group 3 (Active Comparator): BOOI<20, BCI≥ 100 Alfuzosin was administered daily (10 mg) for 12 month.
  Interventions: Drug: Alfuzosin
- group 4 (Active Comparator): BOOI<20, BCI<100 Alfuzosin was administered daily (10 mg) for 12 month.
  Interventions: Drug: Alfuzosin

INTERVENTIONS:
Drug: Alfuzosin — 10mg, once daily, 12months
  Other Names: xatral
  Arms: group1
Drug: Alfuzosin — 10mg, once daily, 12months
  Other Names: xatral
  Arms: group2
Drug: Alfuzosin — 10mg, once daily, 12months
  Other Names: xatral
  Arms: group 3
Drug: Alfuzosin — 10mg, once daily, 12months
  Other Names: xatral
  Arms: group 4

SUMMARY:
Benign prostatic hyperplasia (BPH) is a common condition among older men. The efficacy of α1-blockers for treating BPH has been well documented and they are recommended for the treatment of BPH by clinical guidelines.

It is not well known if a stratification based on the grade of BOO and bladder contractility has any predictive value for patients who are treated with an α1-selective blocking agent. In our study, we investigated possible differences in treatment outcome between patients with and without BOO, and with or without proper contractility who are treated with alfuzosin. So we will compare the quantified improvements 12 months after alfuzosin medication in LUTS/BPH patients by the grade of BOO and/or bladder contractility.

DETAILED DESCRIPTION:
1. Primary objective To evaluate efficacy on voiding and storage symptoms in LUTS/BPH patients after 12 months of treatment with Xatral XL® by the grade of bladder outlet obstruction and/or bladder contractility
2. Secondary objectives To evaluate efficacy on voiding and storage symptoms in LUTS/BPH patients after 3 months and 6 months of treatment with Xatral XL® by the grade of bladder outlet obstruction and/or bladder contractility To evaluate efficacy on maximal flow rate (MFR) and post-voided residual urine (PVR) To evaluate on voiding frequency, urgency severity & frequency, and nocturia To evaluate patient tolerability to the medication To evaluate global impression of improvement (GII)

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory males (≥50 years) suffering from LUTS suggestive of BPH
* Patients satisfying all of the following:
* Moderate to severe LUTS :
* international prostate symptom score (IPSS)≥ 8
* An enlarged prostate (≥25 mL)
* Decreased peak flow rate : Qmax ≤15 mL/s (volume voided ≥ 120 mL)

Exclusion Criteria:

* Post voided residual urine ≥ 200 mL
* Patients performing catheterization
* Urinary tract infection patients
* Patients taking 5 alpha reductase inhibitor
* Known hypersensitivity to alfuzosin
* History of postural hypotension or syncope
* Hypertension patients treated with other alpha1-blockers
* Patients newly taking anticholinergic medication within 1 month
* Hepatic insufficiency (Aspartate transaminase /alanine aminotransferase ≥ 2 times of normal range)
* Renal insufficiency (s-Cr ≥ 2mg/dL)
* Unstable angina pectoris
* Uninvestigated hematuria
* Serum Prostate specific antigen ≥ 4 ng/mL (biopsy proven no cancer patients can be included)
* Interstitial cystitis patients
* Severe concomitant condition threatening life.
* Patient who is unable to make voiding diary
* Bladder or prostate cancer patients
* Patients receiving prostate or bladder surgery

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, M.D., PhD, Principal Investigator — From the Department of Urology, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a specialty clinic at the Asan Medical Center, Samsung Medical Center,The Catholic University of Korea College of Medicine, Hallym University, Chuncheon, Korea for 12-month
Pre-assignment Details: 232 participants recruited; 276 screened, 44 excluded
Groups:
- BOOI≥20, BCI≥ 100: Bladder outlet obstruction index(BOOI)≥ 20, bladder contractility index (BCI)≥ 100
  alfuzosin : 10mg, once daily, 12months
- BOOI≥20, BCI< 100: BOOI≥ 20, BCI<100
  alfuzosin : 10mg, once daily, 12months
- BOOI<20, BCI≥ 100: BOOI<20, BCI≥ 100)
  alfuzosin : 10mg, once daily, 12months
- BOOI<20, BCI< 100: BOOI<20, BCI<100
  alfuzosin : 10mg, once daily, 12 months
Period: Overall Study
Arm/Group | BOOI≥20, BCI≥ 100 | BOOI≥20, BCI< 100 | BOOI<20, BCI≥ 100 | BOOI<20, BCI< 100
Started | 61 | 76 | 41 | 54
Completed | 41 | 50 | 30 | 44
Not Completed | 20 | 26 | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Group 3: BOOI<20, BCI≥ 100)
  alfuzosin : 10mg, once daily, 12months
- Group 4: BOOI<20, BCI<100
  alfuzosin : 10mg, once daily, 12 months
- group1: BOOI≥ 20, BCI≥ 100
  alfuzosin : 10mg, once daily, 12months
- group2: BOOI≥ 20, BCI<100
  alfuzosin : 10mg, once daily, 12months
- Total: Total of all reporting groups
Arm/Group | Group 3 | Group 4 | group1 | group2 | Total
Number analyzed (Participants) | 41 | 54 | 61 | 76 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 31 | 44 | 51 | 66 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (2.0) | 67.4 (0) | 66.0 (1.2) | 63.1 (5) | 65.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 41 | 54 | 61 | 76 | 232
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 41 | 54 | 61 | 76 | 232
international prostate symptom score [Mean (Standard Deviation); unit: scores] — higher values represent a worse outcome total score range (form 0 to 35)
  scores | 18.9 (7.6) | 18.8 (6.8) | 19.4 (6.9) | 21.0 (6.5) | 19.5 (6.95)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome; International Prostate Symptom Score Changes Between 4 Groups Compared to Baseline After 12 mo Treatment
Description: international prostate symptom score was measured at baseline and 12 months. total scores on a scale range (from 0 to 35) higher values represent a worse outcome
  Baseline score minus 12-month score
Time Frame: 12months
Measure: Mean (Standard Deviation); unit: score
Groups:
- BOOI≥ 20, BCI≥100: Bladder outlet obstruction index(BOOI)≥ 20, Bladder contractility index(BCI)≥ 100 Alfuzosin was administered daily (10 mg) for 12 month.
  alfuzosin: 10mg, once daily, 12months
- BOOI≥ 20, BCI<100: BOOI≥ 20, BCI<100 Alfuzosin was administered daily (10 mg) for 12 month.
  alfuzosin: 10mg, once daily, 12months
- BOOI<20, BCI≥ 100: BOOI<20, BCI≥ 100 Alfuzosin was administered daily (10 mg) for 12 month.
  alfuzosin: 10mg, once daily, 12months
- BOOI<20, BCI<100: BOOI<20, BCI<100 Alfuzosin was administered daily (10 mg) for 12 month.
  alfuzosin: 10mg, once daily, 12 months
Arm/Group | BOOI≥ 20, BCI≥100 | BOOI≥ 20, BCI<100 | BOOI<20, BCI≥ 100 | BOOI<20, BCI<100
Number analyzed (Participants) | 41 | 50 | 30 | 44
score | 13.0 (6.6) | 12.0 (5.4) | 10.6 (6.1) | 13.4 (6.3)
Statistical Analysis 1: Comparison: BOOI≥ 20, BCI≥100 vs BOOI≥ 20, BCI<100 vs BOOI<20, BCI≥ 100 vs BOOI<20, BCI<100; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

2. Primary Outcome: Treatment Efficacy Was Analyzed by Validated Symptom Scores.
Description: Alfuzosin was administered daily (10 mg). After 12 months of treatment, efficacy and safety were analyzed. Efficacy was measured by validated symptom scores (using IPSS ). IPSS score change was measured pre- and post- treatment.
Time Frame: 12 month
Population: The population analyzed included participants receiving drug for 12 months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Group 3 | Group 4 | group1 | group2
Number analyzed (Participants) | 30 | 44 | 41 | 50
score | 8.3 (6.2) | 6.4 (6.2) | 6.4 (6.5) | 9.0 (6.1)
Statistical Analysis 1: Comparison: Group 3 vs Group 4 vs group1 vs group2; The Kruskal-Wallis test, analysis of variance, and the Wilcoxon signed rank-sum test were used to compare changes from baseline to endpoint after treatment; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

3. Secondary Outcome: Changes of International Continence Society (ICS)-Male Questionnaire (Voiding Sum)
Description: Changes of International Continence Society (ICS)-male questionnaire (voiding sum) to measure the efficacy of alfuzosin 10mg at 12 months post-treatment.
  Range 0-20, higher scores represent worse outcomes.
Time Frame: 12months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | group1 | group2 | Group 3 | Group 4
Number analyzed (Participants) | 41 | 50 | 30 | 44
score on a scale | 8.2 (4.3) | 7.2 (3.4) | 9.7 (6.4) | 8.2 (4.1)

4. Secondary Outcome: Changes of Peak Flow Rates on Uroflowmetry
Description: Changes of peak flow rates on uroflowmetry to measure the efficacy of alfuzosin 10mg at 12 months post-treatment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | group1 | group2 | Group 3 | Group 4
Number analyzed (Participants) | 41 | 50 | 30 | 44
ml/s | 14.3 (7.2) | 10.9 (6.4) | 16.8 (8.7) | 13.0 (5.3)

5. Secondary Outcome: Changes in Residual Urine Volumes
Description: Changes in residual urine volumes to measure the efficacy of alfuzosin 10mg at 12 months post-treatment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | group1 | group2 | Group 3 | Group 4
Number analyzed (Participants) | 41 | 50 | 30 | 44
ml | 51.6 (87) | 37 (45.2) | 29.3 (35.9) | 31.7 (35.3)

ADVERSE EVENTS:
Arm/Group | Group 3 | Group 4 | group1 | group2
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/54 | 0/61 | 0/76
Other Adverse Events (participants affected / at risk) | 2/41 | 2/54 | 2/61 | 3/76
OTHER ADVERSE EVENTS (reported when occurring in more than 3.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 3 (N=41) | Group 4 (N=54) | group1 (N=61) | group2 (N=76)
dizziness (Vascular disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Patients were not divided into three groups according to the ICS nomogram (obstructed [BOOI <40], equivocally obstructed (20 <BOOI <40), and unobstructed [BOOI <20]).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes